CLINICAL TRIAL: NCT00371150
Title: A Study to Describe the Antiviral Effect of Entecavir (ETV) in Blacks/African Americans and Hispanics With Chronic Hepatitis B Virus (HBV) Infection Who Are Nucleoside-Naive
Brief Title: Effect of Entecavir in Blacks/African Americans and Hispanics With Chronic Hepatitis B Virus (HBV) Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI463-085
Record Dates: First submitted 2006-08-29; First posted 2006-09-01 (Estimated); Results first posted 2012-04-16 (Estimated); Last update posted 2012-04-16 (Estimated); Status verified 2012-03

CONDITIONS: Hepatitis B Infection
MeSH Terms: conditions — Hepatitis B | interventions — entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm1 (Experimental)
  Interventions: Drug: Entecavir

INTERVENTIONS:
Drug: Entecavir — Tablets, Oral, 0.5 mg, once daily, up to 52 weeks
  Other Names: Baraclude; BMS-200475

SUMMARY:
The purpose of this clinical research study is to develop observational clinical experience with the use of entecavir in participants who are either of Black/African-American race or of Hispanic ethnicity.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HBV infection, with either HBeAg-positive (HBeAb-negative) or HBeAg-negative (HBeAb-positive) disease
* Black/African American Race and/or Hispanic ethnicity
* Nucleoside/tide-naive
* Males or females ≥ 16 years of age (or minimum age required in a given country)
* Compensated liver function
* ALT of 1.3 to 10 x upper limit of normal (ULN)
* No Co-infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV) or hepatitis D virus (HDV)

Exclusion Criteria

* Women of childbearing potential (WOCBP) who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 6 weeks after study medication has been discontinued
* Women who are pregnant or breastfeeding
* Women with a positive pregnancy test on enrollment or prior to study drug administration
* Evidence of decompensated cirrhosis including but not limited to: variceal bleeding; hepatic encephalopathy; or ascites requiring management with diuretics or paracentesis
* Recent history of pancreatitis (resolution of any recent pancreatitis must be documented by normal lipase at least 12 weeks prior to the first dose of study medication)
* Currently abusing illegal drugs or alcohol sufficient, in the investigator's opinion, to prevent adequate compliance with study therapy or to increase the risk of hepatotoxicity or pancreatitis
* Other serious medical conditions that might preclude completion of this study or that require chronic administration of prohibited medications
* Serum creatinine > 1.5 mg/dL
* Hemoglobin < 10.0 g/dL
* Platelet count < 70,000/mm3
* Absolute neutrophil count < 1200 cells/mm3
* Serum alpha fetoprotein (AFP) level > 100 ng/mL. If the AFP level is between 21 and 100 ng/mL, it must be repeated. If the repeat AFP level is between 21 and 100 ng/mL and if ultrasonography or computerized tomography (CT) of the liver performed prior to the first dose of study medication does not demonstrate a focal lesion suggestive of carcinoma, the subject may be dosed in the study
* Known history of allergy to nucleoside analogues
* Any prior therapy with Entecavir
* Any prior or concomitant use of nucleoside or nucleotide analogue antiviral agents with activity against hepatitis B (e.g., ETV, lamivudine (LVD), tenofovir [TDF], emtricitabine (FTC), clevudine, telbivudine [LdT], famciclovir), or any other experimental anti-HBV antiviral agent
* Therapy with interferon, thymosin alpha or other immunostimulators within 24 weeks of enrollment (i.e., dosing) into this study
* Subjects who require chronic administration of concomitant medications which cause immunosuppression or which are associated with a high rate of nephrotoxicity or hepatotoxicity, or which affect renal excretion, should not be enrolled in this study
* Unable to tolerate oral medication
* Poor peripheral venous access
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled into this study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2006-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (25):
- United States (14):
  - Alabama Liver & Digestive Specialists (Alds), Montgomery, Alabama
  - University Of Arizona, Tucson, Arizona
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - University Of Miami, Miami, Florida
  - Empire International Research, Miami, Florida
  - University Of Chicago, Chicago, Illinois
  - Banks Hepatology Institute, Pc, College Park, Maryland
  - Brigham And Women'S Hospital, Boston, Massachusetts
  - L L C Bda The Research Institute, Springfield, Massachusetts
  - Va New York Harbor Healthcare System, New York, New York
  - Westchester Digestive Disease Group, Llp, Yonkers, New York
  - Albert Einstein Healthcare Network, Philadelphia, Pennsylvania
  - Alamo Medical Research, San Antonio, Texas
  - Hunter Holmes Mcguire D V A M C, Richmond, Virginia
- Brazil (5):
  - Local Institution, Salvador, Estado de Bahia
  - Local Institution, Belo Horizonte - Mg, Minas Gerais
  - Local Institution, Rio de Janeiro - Rj, Rio de Janeiro
  - Local Institution, Campinas, São Paulo
  - Local Institution, Sao Paulo - Sp, São Paulo
- Mexico (3):
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Zapopan, Jalisco
  - Local Institution, Df, Mexico City
- Local Institution, Santurce, Puerto Rico
- South Africa (2):
  - Local Institution, Belville, Western Cape
  - Local Institution, Goodwood, Western Cape

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 131 participants were enrolled at 27 sites.
Pre-assignment Details: Of the 131 participants enrolled, 85 were never treated (82 no longer met study criteria, 2 withdrew consent, and 1 had other reason).
Groups:
- Black/ African American: Entecavir (ETV) tablets, Oral, 0.5 mg, once daily, up to 52 weeks
- Hispanic: ETV tablets, Oral, 0.5 mg, once daily, up to 52 weeks
Period: Overall Study
Arm/Group | Black/ African American | Hispanic
Started | 40 | 6
Discontinued Prior to Week 48 Visit | 1 | 1
Discontinued at or After Week 48 Visit | 2 | 1
Completed | 37 ("Completion of treatment" means received treatment through Week 52) | 4 ("Completion of treatment" means received treatment through Week 52)
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Black/ African American | Hispanic | Total
Number analyzed (Participants) | 40 | 6 | 46
Age Continuous [Median (Full Range); unit: years] | 39.0 [22 to 67] | 48.0 [29 to 69] | 40.0 [22 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 2 | 11
  Male | 31 | 4 | 35
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic / Latino | 0 | 6 | 6
  Not Hispanic / Latino | 18 | 0 | 18
  Missing | 22 | 0 | 22
Race/Ethnicity, Customized [Number; unit: participants]
  Black/ African American | 40 | 0 | 40
  White | 0 | 6 | 6
Region of Enrollment [Number; unit: participants]
  Brazil | 21 | 0 | 21
  Mexico | 0 | 2 | 2
  South Africa | 3 | 0 | 3
  United States | 16 | 4 | 20
Hepatitis B surface antigen (HBsAg) status at baseline [Number; unit: participants]
  Positive | 40 | 4 | 44
  Negative | 0 | 0 | 0
  Missing | 0 | 2 | 2
Hepatitis B e antigen (HBeAg) status at baseline [Number; unit: participants]
  Positive | 22 | 4 | 26
  Negative | 18 | 2 | 20
Hepatitis B e antibody (HBeAb) at baseline [Number; unit: participants]
  Positive | 19 | 2 | 21
  Negative | 21 | 4 | 25
Alanine Aminotransferase (ALT) [Median (Full Range); unit: U/L] | 106 [30 to 617] | 113 [80 to 301] | 107 [30 to 617]
Albumin [Median (Full Range); unit: g/dL] | 4.3 [3.0 to 5.1] | 4.3 [3.5 to 4.6] | 4.3 [3.0 to 5.1]
Total Bilirubin [Median (Full Range); unit: mg/dL] | 0.6 [0.3 to 2.1] | 0.5 [0.3 to 1.1] | 0.6 [0.3 to 2.1]

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants Who Achieve HBV DNA < Lower Limit of Quantitation (LOQ = 29 IU/mL [Approximately 169 Copies/mL]) at Week 48
Description: HBV DNA assessments were performed using the Roche COBAS® TaqMan AmpliPrep assay. LOQ is the level above which quantitative results may be obtained with a specified degree of confidence. The LOQ is mathematically defined as equal to 10 times the standard deviation of the results for a series of replicates used to determine a justifiable limit of detection.
Time Frame: Week 48
Population: All treated participants. If a participant is missing the efficacy assessments for a visit, this is considered a failure and is counted as evaluable.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Black / African American: ETV tablets, Oral, 0.5 mg, once daily, up to 52 weeks
- Total: ETV tablets, Oral, 0.5 mg, once daily, up to 52 weeks (Includes 6 participants of the Hispanic cohort)
Arm/Group | Black / African American | Total
Number analyzed (Participants) | 40 | 46
percentage of participants | 12.5 [NA to NA] — Since enough participants could not be enrolled in the Hispanic cohort, 95% CI analysis was only performed on the overall population. | 13.0 [3.3 to 22.8]

2. Secondary Outcome: Percentage of Participants With HBV DNA by PCR Category at Week 48
Description: HBV DNA assessments were performed using the Roche COBAS® TaqMan AmpliPrep assay.
Time Frame: Week 48
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Black / African American | Total
Number analyzed (Participants) | 40 | 46
percentage of participants
  <50 IU/mL (< 300 copies/mL) | 72.5 | 69.6
  50 to <172 IU/mL (300 to < 103 copies/mL) | 0 | 0
  172 to <1720 IU/mL (103 to < 104 copies/mL) | 10.0 | 10.9
  1720 to <17200 IU/mL (104 to < 105 copies/mL) | 5.0 | 4.3
  ≥17,200 IU/mL (≥105 copies/mL) | 0 | 0
  Missing | 12.5 | 15.2

3. Secondary Outcome: Percentage of Participants With Virologic Rebound Through Week 48 While on Continued Dosing With ETV
Description: Virologic rebound is defined as a confirmed increase of ≥ 1 log10 in HBV DNA from the participant's nadir value (2 sequential HBV DNA measurements or last on-treatment measurement)
Time Frame: through Week 48
Population: All treated participants. The participants who discontinued prior to Week 48 were counted as failure.
Measure: Number; unit: percentage of participants
Arm/Group | Black / African American | Total
Number analyzed (Participants) | 40 | 46
percentage of participants | 0 | 0

4. Secondary Outcome: Percentage of Participants With Alanine Aminotransferase (ALT) Normalization at Week 48
Description: ALT normalization=ALT level being less than or equal to 1 times the upper limit of normal (ULN). ULN for ALT is 37 U/L.
Time Frame: Week 48
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Black / African American | Total
Number analyzed (Participants) | 40 | 46
percentage of participants | 67.5 | 67.4

5. Secondary Outcome: Percentage of Participants With Confirmed HBeAg Loss at Week 48 (for HBeAg-positive Participants Only)
Description: HBeAg is a hepatitis B viral protein. HBeAg loss = HBeAg-negative at the specified analysis week
Time Frame: Week 48
Population: Treated HBeAg-positive participants. If a participant was missing the efficacy assessments for a visit, this is considered a failure and was counted as evaluable.
Measure: Number; unit: percentage of participants
Arm/Group | Black / African American | Total
Number analyzed (Participants) | 22 | 26
percentage of participants | 50.0 | 53.8

6. Secondary Outcome: Percentage of Participants With HBeAg Seroconversion at Week 48 (for HBeAg-positive Participants Only)
Description: HBeAg is a hepatitis B viral protein. HBeAg Seroconversion = HBeAg Loss and Presence of Hepatitis B e Antibody (HBeAb).
Time Frame: Week 48
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Black / African American | Total
Number analyzed (Participants) | 22 | 26
percentage of participants | 40.9 | 46.2

7. Secondary Outcome: Percentage of Participants With Hepatitis B Surface Antigen (HBsAg) Loss at Week 48
Description: HBsAg = a part of the hepatitis B virus that, when in the blood, is a marker of infection. HBsAg loss = HBsAg-negative at the specified analysis week.
Time Frame: Week 48
Population: All treated participants. If a participant was missing the efficacy assessments for a visit, this is considered a failure and was counted as evaluable.
Measure: Number; unit: percentage of participants
Arm/Group | Black / African American | Total
Number analyzed (Participants) | 40 | 46
percentage of participants | 5.0 | 6.5

8. Secondary Outcome: Percentage of Participants With HBsAg Seroconversion at Week 48
Description: HBsAg = a part of the hepatitis B virus that, when in the blood, is a of infection. HBs seroconversion is defined as HBsAg loss with positive HBsAb.
Time Frame: Week 48
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Black / African American | Total
Number analyzed (Participants) | 40 | 46
percentage of participants | 2.5 | 4.3

9. Secondary Outcome: Mean log10 Reduction From Baseline in HBV DNA at Week 48
Description: HBV DNA was analyzed by PCR, using the Roche COBAS®TaqMan TaqMan AmpliPrep assay. Reduction in log10 HBV count=reduced viral load.
Time Frame: baseline, Week 48
Population: All treated participants. The participants who discontinued prior to Week 48 were counted as failure.
Measure: Mean (Standard Error); unit: log10 IU/mL
Arm/Group | Black / African American | Total
Number analyzed (Participants) | 35 | 39
log10 IU/mL
  Baseline | 7.1 (0.26) | 7.0 (0.25)
  HBV DNA at Week 48 | 1.88 (0.100) | 1.87 (0.091)
  Change from baseline | -5.22 (0.249) | -5.18 (0.231)

10. Secondary Outcome: Percentage of Participants With HBV DNA < Other IU Cut-off Points That May be Clinically Relevant at the Time of Data Analysis
Time Frame: Week 48
Population: Since there were no other cut-off points other than those at the time of data analysis, this outcome was not analysed.
Measure: Number; unit: percentage of participants
Groups:
- Black / African American; Total: Entecavir tablets, Oral, 0.5 mg, once daily, up to 52 weeks
Arm/Group | Black / African American | Total
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Number of Participants With Adverse Events (AE), Serious Adverse Events (SAE), and Discontinuations From Study Drug Due to Adverse Events
Description: AE: any new untoward medical occurrence/worsening of pre-existing medical condition, whether or not related to study drug. SAE: any AE that resulted in death; was life threatening; resulted in persistent/significant disability/incapacity; resulted in/prolonged an existing in-patient hospitalization; was a congenital anomaly/birth defect; or was an overdose. Participants who discontinued the study due to any AEs were recorded.
Time Frame: From enrollment through Week 52 + 5 days
Population: All treated participants.
Measure: Number; unit: participants
Groups:
- Hispanic; Total: Entecavir tablets, Oral, 0.5 mg, once daily, up to 52 weeks
Arm/Group | Black / African American | Hispanic | Total
Number analyzed (Participants) | 40 | 6 | 46
participants
  Deaths | 0 | 0 | 0
  SAEs | 3 | 1 | 4
  Discontinuations Due to AEs | 0 | 0 | 0
  Any AE | 33 | 5 | 38
  Grade 3 - 4 AEs | 5 | 1 | 6
  Related AEs | 16 | 0 | 16
  Grade 2 - 4 Related AEs | 5 | 0 | 5

12. Secondary Outcome: Number of Participants With Laboratory Abnormalities On-treatment (OT) and Off-Treatment (OF): Hematology
Description: Criteria for hematology abnormalities were graded using the modified WHO grading system. Hemoglobin: <=11.0 g/dL; White Blood Cells: <4000/mm^3; Absolute Neutrophils (includes absolute bands): <1500/mm^3; Platelets: <=99,000/mm^3; International Normalized Ratio: ≥ 1.5 and ≥ 0.5 from baseline.
Time Frame: OT: From start of study therapy through Week 52 + 5 days; OF= End of OT period + 24-week follow-up
Population: All treated participants. n = number of participants in the OF period.
Measure: Number; unit: participants
Groups:
- Total: Entecavir tablets, Oral, 0.5 mg, once daily, up to 52 weeks (Includes 6 participants of the Hispanic cohort)
Arm/Group | Black / African American | Total
Number analyzed (Participants) | 40 | 46
participants
  Hemoglobin-OT | 1 | 2
  Hemoglobin-OF; n=26 , 29 | 0 | 0
  White Blood Cells-OT | 15 | 18
  White Blood Cells-OF; n=26 , 29 | 7 | 8
  Neutrophils -OT | 13 | 13
  Neutrophils-OF; n=26 , 26 | 4 | 4
  Platelets-OT | 4 | 4
  Platelets-OF; n=26 , 29 | 0 | 0
  International Normalized Ratio-OT | 18 | 23
  International Normalized Ratio-OF; n=26 , 29 | 4 | 4

13. Primary Outcome: Percentage of Participants With HBV Deoxyribonucleic Acid (DNA) < 50 IU/mL by Polymerase Chain Reaction (PCR) at Week 48
Description: HBV DNA assessments were performed using the Roche COBAS® TaqMan AmpliPrep assay. HBV DNA < 50 IU/mL = approximately <300 copies/mL.
Time Frame: Week 48 of ETV treatment
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Black / African American | Total
Number analyzed (Participants) | 40 | 46
percentage of participants | 72.5 [NA to NA] — Since enough participants could not be enrolled in the Hispanic cohort, 95% CI analysis was only performed on the overall population. | 69.6 [56.3 to 82.9]

14. Secondary Outcome: Number of Participants With Laboratory Abnormalities On-treatment (OT) and Off-Treatment (OF) : Serum Chemistry
Description: The modified World Health Oranization(WHO)grading system was used to grade the abnormalities. ULN=upper limit of normal. Alanine aminotransferase:>1.25xULN, Aspartate aminotransferase:>1.25xULN, Alkaline Phosphatase:>1.25xULN, Total Bilirubin:>1.1xULN, Serum Lipase:>1.10xULN, Creatinine:>1.1xULN, Blood Urea Nitrogen:1.25xULN, Hyperglycemia:>116 mg/dL, Hypoglycemia:<64 mg/dL, Hyponatremia:<132meq/L, Hypokalemia:<3.4 meq/L, Albumin:≥1g/dL decrease from baseline, <3 g/dL; Hypernatremia:>148 meq/L, Hyperkalemia:>5.6 meq/L, Hypokalemia:<3.4 meq/L, Hyperchloremia:>113 meq/L, Hypochloremia:<93 meq/L
Time Frame: OT: From start of study therapy through Week 52 + 5 days; OF= End of OT period + 24-week follow-up
Population: All treated participants. n = number of participants in the OF period.
Measure: Number; unit: participants
Arm/Group | Black / African American | Total
Number analyzed (Participants) | 40 | 46
participants
  Alanine aminotransferase-OT | 37 | 43
  Alanine aminotransferase-OF; n=26 , 29 | 3 | 4
  Aspartate aminotransferase-OT | 33 | 38
  Aspartate aminotransferase-OF; n=26 , 29 | 2 | 3
  Alkaline Phosphatase-OT | 3 | 3
  Alkaline Phosphatase-OF; n=26 , 29 | 1 | 1
  Albumin-OT | 3 | 5
  Albumin-OF; n=26 , 29 | 0 | 0
  Total Bilirubin-OT | 7 | 7
  Total Bilirubin-OF; n=26 , 29 | 3 | 4
  Serum Lipase-OT | 12 | 14
  Serum Lipase-OF; n=26 , 29 | 1 | 1
  Creatinine-OT | 3 | 3
  Creatinine-OF; n=26 , 29 | 0 | 0
  Blood Urea Nitrogen-OT | 2 | 2
  Blood Urea Nitrogen-OF; n=26 , 29 | 0 | 0
  Hyperglycemia-OT | 14 | 15
  Hyperglycemia-OF; n=26 , 29 | 5 | 5
  Hypoglycemia-OT | 5 | 5
  Hypoglycemia-OF; n=26 , 29 | 1 | 1
  Hypernatremia-OT | 0 | 0
  Hypernatremia-OF; n=26 , 29 | 0 | 0
  Hyponatremia-OT | 3 | 3
  Hyponatremia-OF; n=26 , 29 | 0 | 1
  Hyperkalemia-OT | 0 | 0
  Hyperkalemia-OF; n=26 , 29 | 0 | 0
  Hypokalemia-OT | 3 | 3
  Hypokalemia-OF; n=26 , 29 | 0 | 0
  Hyperchloremia-OT | 0 | 0
  Hyperchloremia-OF; n=26 , 29 | 0 | 0
  Hypochloremia-OT | 0 | 0
  Hypochloremia-OF; n=26 , 29 | 0 | 0

ADVERSE EVENTS:
Time Frame: 52 Weeks
Groups:
- Entecavir (ETV): Entecavir tablets, Oral, 0.5 mg, once daily, up to 48 weeks (Includes 6 participants of the Hispanic cohort)
Arm/Group | Entecavir (ETV)
Serious Adverse Events (participants affected / at risk) | 4/46
Other Adverse Events (participants affected / at risk) | 21/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Entecavir (ETV) (N=46)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
PYREXIA (General disorders) | 1
ANGINA PECTORIS (Cardiac disorders) | 1
ASCITES (Gastrointestinal disorders) | 1
BLOOD GLUCOSE ABNORMAL (Investigations) | 1
HEADACHE (Nervous system disorders) | 1
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1
LOBAR PNEUMONIA (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Entecavir (ETV) (N=46)
SOMNOLENCE (Nervous system disorders) | 3
PYREXIA (General disorders) | 4
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4
HEADACHE (Nervous system disorders) | 8
URINARY TRACT INFECTION (Infections and infestations) | 3
ABDOMINAL PAIN (Gastrointestinal disorders) | 6
DIARRHOEA (Gastrointestinal disorders) | 5
FATIGUE (General disorders) | 4
MYALGIA (Musculoskeletal and connective tissue disorders) | 3
NASOPHARYNGITIS (Infections and infestations) | 3
INFLUENZA (Infections and infestations) | 4
NAUSEA (Gastrointestinal disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication